CLINICAL TRIAL: NCT02171338
Title: Procalcitonin as a Marker of Antibiotic Therapy in Patients With Lower Respiratory Tract Infections. Can Measurement of Procalcitonin Reduce the Use of Antibiotics?
Brief Title: Procalcitonin as a Marker of Antibiotic Therapy in Patients With Lower Respiratory Tract Infections
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Holbaek Sygehus (Other)
Collaborators: Region Sjælland (Other); Aase and Ejnar Danielsens Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SJ-342; SJ-RO-01, j.nr. 12-000179 (Registry Identifier: Region Sjaelland, Datatilsynet)
Record Dates: First submitted 2014-06-17; First posted 2014-06-24 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Pneumonia; Acute Exacerbation of Chronic Obstructive Airways Disease
Keywords: Procalcitonin; Antibiotic therapy; Lower respiratory tract diseases
MeSH Terms: conditions — Pneumonia | interventions — Moxifloxacin; Azithromycin; Penicillin G; Cefuroxime; Ciprofloxacin; Clarithromycin; Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotic treatment based on PCT-level (Other): Information regarding the PCT-levels in the intervention group is available to the treating doctor and the test subjects are randomized for treatment based on the level of PCT (PCT algorithm).
  With a PCT ≥0.25 µg/l and ≥0.10 µg/l for pneumonia and AECOPD respectively antibiotic treatment is advised to be started.
  Interventions: Other: PCT-level; Behavioral: Antibiotic treatment based on PCT-level
- Control (No Intervention): Test subjects randomized for standard treatment (control group) are treated in accordance with the existing treatment guidelines of Holbaek Hospital.
  PCT-level will be measured but the treating doctor has no access to the result.

INTERVENTIONS:
Other: PCT-level — PCT-level is available to the treating doctor.
  Arms: Antibiotic treatment based on PCT-level
Behavioral: Antibiotic treatment based on PCT-level — PCT-level is available to the treating doctor and the decision whether or not to treat with antibiotic is based on the level of PCT.
  The type of antibiotic chosen to treat is based on the existing antibiotic treatment guidelines of Holbaek Hospital and includes the antibiotics listed above.
  Other Names: Avelox®; Azithromycin; Benzylpenicillin; Bioclavid®; Cefuroxim; Ciprofloxacin; Clarithromycin; Piperacillin/Tazobactam; Primcillin; Vepicombin®; Zinacef®
  Arms: Antibiotic treatment based on PCT-level

SUMMARY:
The purpose of this study is to investigate weather or not the use of a procalcitonin(PCT)-based treatment in the daily clinical work could lower the consumption of antibiotics in patients with lower respiratory tract infections.

DETAILED DESCRIPTION:
An increasing amount of antibiotics are being consumed and along with the increased resistance they carry along, they pose an increasing problem for the health sector. A method to decrease the use of antibiotics is highly desirable and of great importance in order to halt the spread of multi-resistant bacteria that is becoming an increasing problem in Denmark.

Lower respiratory tract infections such as pneumonia and acute exacerbations of chronic obstructive pulmonary disease (AECOPD) are frequent reasons for patient contact in both the primary and secondary sectors. Identifying which patients that could benefit from treatment with antibiotics is a great challenge to the health sector. This is why patients often are treated with antibiotics if there is a mere suspicion of the above-mentioned disorders, even if they are not proved for certain.

An increasing amount of data suggests that procalcitonin (PCT) could serve as a possible marker of respiratory tract infections caused by bacteria. Alongside the conventional clinical parameters, the level of PCT is regarded as a promising means to decide whether to treat with antibiotics and how long such a treatment should endure. When an infection is under control by the immune system of the individual or by treatment with antibiotics, the level of PCT will diminish by 50% on a daily basis. Accordingly, a decline in the PCT levels should indicate a favorable response to antibiotic treatment. Therefore there is a need to further investigate if the PCT levels can be used, in the everyday clinic, to diagnose patients with pneumonia or AECOPD caused by bacteria and if this could have an effect on the use of antibiotics, thus optimizing the treatment of the patients.

The purpose of this research project is to compare the amount of antibiotics consumed using standard treatment and treatment based on the PCT levels of patients with lower respiratory tract infections, respectively.

With the research at hand, a clarification of whether a measurement of PCT can serve as a diagnostic tool to distinguish between bacterial and non-bacterial infections in patients that are suspected of having pneumonia or AECOPD is desirable. In extension, this study wants to clarify if the PCT levels can indicate when a potential antibiotic treatment should be initiated and if the use of a PCT-based treatment in the daily clinical work could lower the consumption of antibiotics.

The hypothesis is that PCT will be increased (≥0.25 µg/l and ≥0.10 µg/l for pneumonia and AECOPD respectively) in lower respiratory tract infections caused by bacteria, whereas PCT should only be slightly increased in non-bacterial lower respiratory tract infections if at all. It is expected that using a PCT-based treatment in lower respiratory tract infections could lower the consumption of antibiotics, while at the same time it should not prove a greater health risk to patients than by using a standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in Holbæk Hospital
* Clinical and paraclinical signs of pneumonia and/or AECOPD.

Exclusion Criteria:

* Unable to hand over written consent.
* Terminal patients.
* Patients with known abscess in the lungs and/or emphysema.
* Patients who have received treatment with strong doses (>5mg/day) of biotin (vitamin B7 og B8) within the last eight hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-08 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Days of antibiotic treatment | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks, and up to 2 weeks after discharge.

SECONDARY OUTCOMES:
Numbers of days admitted | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
  Numbers of days admitted from the day og enrollment in the study to the day of discharge.

OTHER OUTCOMES:
Patients with low PCT-level | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.
  Numbers of patients with a PCT-level ≤0,1 µm/L and ≤0,25 µm/L in AECOPD and pneumonia respectively who gets treated with antibiotics during their hospitalization.
Recurrence within 30 days after discharge | From 1 to 30 days after discharge
  Numbers of patients with recurrence of AECOPD or pneumonia within 30 days after discharge.
Type of antibiotics | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks, and up to 2 weeks after discharge.
  Antibiotics used to treat the enrolled patients (name, i.v. or p.o.)
Death and adverse events in the two treatment groups | Participants will be followed for the duration of hospital stay, an expected average of 2 weeks, and up to 30 days after discharge.
  Death and adverse events in the two treatment groups meaning:
  * Death by any cause
  * Complications in connection with lower respiratory tract infections (empyema, abscess)
  * Severe complications from treatment with antibiotics (anaphylactic shock, rash)
  * Admission to intensive care unit
  * Readmission within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Hans Ibsen, M.D., D.M.Sc, Study Director — Holbaek Sygehus
Locations (1):
- Holbæk Hospital, Holbæk, Holbæk, Denmark